CLINICAL TRIAL: NCT04866875
Title: Impact of Different Rates of Weight Loss on Final Outcomes in Pre-menopausal Women
Brief Title: Investigating the Early Markers of Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Eric Doucet, Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMRU
Record Dates: First submitted 2018-10-09; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Weight Loss; Appetitive Behavior; Obesity
Keywords: energy expenditure; weight loss; appetite; impulsivity; food reward
MeSH Terms: conditions — Weight Loss; Appetitive Behavior; Obesity; Impulsive Behavior | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid weight loss (Active Comparator): Participants in this group will be deprived in 1000 kcal/day (calculated based on their individual energy requirements) for 10 weeks
  Interventions: Behavioral: dieting
- Slow weight loss (Experimental): Participants in this group will be deprived in 500 kcal/day (calculated based on their individual energy requirements) for 20 weeks
  Interventions: Behavioral: dieting

INTERVENTIONS:
Behavioral: dieting — The minimum amount of caloric intake will be pre-set in 1200 kcal for the both groups, in order to avoid micronutrient deficiencies during the intervention. The diet macronutrient composition will be personalized for each participant based on the results of 2-day energy intake at preliminary session, measured with food items selected from a validated food menu. Individuals will be instructed to maintain the level of energy restriction and macronutrient composition during the diet period, however they will be able to do food exchanges, based on the Canadian Diabetes Association system . This method allows individuals to select foods they enjoy during the weight loss, however in smaller quantities.
  Other Names: Caloric restriction (-500 kcal/day); Caloric restriction (-1000 kcal/day)

SUMMARY:
The study will include 30 women randomized in two distinct groups: G1: Slow weight loss and G2: Rapid weight loss . The total duration of the program will be different for each group, being over 20 and 10 weeks for G1 and G2, respectively, in attempt to match the groups on amount of weight loss (approximately 20 pounds per subject). Participants who meet the inclusion criteria will be randomized to rapid or slow weight loss groups. The energy deprivation of the rapid and slow weight loss will be in -1000 kcal/day and -500 kcal/day, respectively. Calculated based on the baseline resting energy expenditure (REE; determined by indirect calorimetry) and their physical activity level measured for one week. The diet macronutrient composition will be personalized for each participant based on the results of 2-day energy intake at preliminary session, measured with food items selected from a validated food menu. Individuals will be instructed to maintain the level of energy restriction and macronutrient composition during the diet period, however they will be able to do food exchanges, based on the Canadian Diabetes Association system. It will be measured participant's body weight, body compositions, appetite sensations, resting energy expenditure, energy intake, palatability, olfactory performance, food reward, food reinforcement and impulsivity. Participants will have 7 sessions in total: 1 preliminary, baseline, 7 days of intervention, 3 follow ups and final assessment.

DETAILED DESCRIPTION:
Preliminary session (approximately 3 hours) During this visit, participants will receive the consent form and they will be informed of the experimental procedures, which will be used during each experimental session, as well as the equipment that will be used to obtain the necessary data. Their weight (digital scale), height (standard stadiometer), waist circumference and blood pressure will be measured at the start the session. If participants match the study inclusion criteria, they will have an equal chance of being assigned to one of two groups; one intervention will last 10 weeks and the second intervention will last 20 weeks but both groups are designed to produce the same amount of weight loss. We will measure their resting metabolism (the energy you use while at rest) (indirect calorimetry). We will then serve a breakfast according to their personal choice and we will recommend them to "eat as much or as little as they want" in 15 minutes. Then, they will be asked to complete other questionnaires the Yale Food Addition Questionnaire that measure personality traits and food addiction symptoms, respectively. This session will be used to determine their breakfast during the experimental sessions and to determine the macronutrient composition (percentage of carbohydrates, fat and protein) will be adopted for them during their diet. They will be asked to fill a food menu and choose your meals for the rest of your day as well as for the day that will follow their visit. We will provide all your food items in lunch boxes and individual bags. They will be able to carry these items and they will be instructed to eat only the items that they have chosen for these 2 days. Lastly, they will be asked to wear a biaxial accelerometer around your upper arm, 24 hours per day during 7 days, including when sleeping, but should remove it when in contact with water (for instance, when bathing, showering or swimming) because this device is not waterproof.

Second Visit: (approximately 1 hour) Upon completion of the preliminary phase, participants will be invited to a 2nd meeting at the lab, in order to receive the dietary instructions related to their weight loss program. This diet is the one that you will be instructed to follow for the duration of the weight loss program (10 or 20 weeks depending on their group). The diet will be prescribed using the Canadian Food Exchange System. This method will allow you to select foods you enjoy during the weight loss, however in smaller quantities.

Exchange lists are groups of foods that contain a similar mix of carbohydrates, protein, fat, and calories. The Canadian exchange system there are seven exchange groups: Grains & Starches; Fruits; Milk & Alternatives; Vegetables; Meat & Alternatives; Fats; Unlimited consumption.

Within any group, participants can exchange one food serving for another. For example, in the Meats group, some sample foods that equal one lean meat exchange might be: 1 oz. of white meat chicken or turkey with no skin or 1 oz. of lean beef.

The daily meal plan will contain foods from all seven Food Exchange lists in order to assure them a complete and a balanced nutrition. However, the number of portions from each group will be recommended based on their individual diet evaluated in the preliminary session. This session will also be used to clarify any potential questions that participants have regarding the project and the intervention.

Third and Fourth experimental sessions (approximately 6 hours each)

Arrival at the laboratory (12 hours fasted, at 7:30 h)

Participants will have a total of 3 experimental sessions: before starting the diet (baseline measurement), 5 to 7 days after the beginning of the weight loss program and at the end of the weight loss program. Each of these visits will take approximately 6 hours. Here is a detailed description of the different methods/procedures that will be employed during each experimental session:

A. Anthropometric, body composition and resting metabolic rate assessments, consumption of a standard breakfast and appetite measurements (Approximately 4.5 hours)-Participant's height and body weight will be measured as soon as they arrive in the laboratory for the experimental session. Their amount of body fat and muscle (by dual energy X-ray absorptiometry) and your resting metabolism (by indirect calorimetry) will also be measured. Afterwards, we will serve breakfast to them. This meal will contain the exact amounts of each item that you consumed during the preliminary session. They will have 15 minutes to consume this entire meal. Additionally, they will be asked to answer 4 specific questions that quantify appetite sensations (desire to eat, hunger, fullness and prospective food consumption) using 100-millimeter visual analogue scales that will be administered before, immediately after (time 0), and every 30 minutes for 3 hours (30, 60, 90, 120, 150 and 180 minutes) following breakfast consumption.

B. Dual energy X-ray absorptiometry (Approximately 10 minutes): We will assess participant's body fat using the dual energy X-ray absorptiometry (DXA). They will be asked to wear a standard issue hospital gown, to lie on an examination table and do not make any movement during the assessment. In the meantime, a low-intensity X-ray will scan your entire body.

C. Indirect Calorimetry (Approximately 45 minutes) - Participant's will be required to remain resting for 30-min during this measurement. A plexiglass hood (similar to a plastic bubble) will be placed over their head through which fresh air will be drawn. The expired air will be sampled for analysis and percentages of oxygen and carbon dioxide will be determined over the 30-min collection period. With this measurement, we will be able to determine participant's resting rate of oxygen consumption. With this information we can calculate their resting rate of energy expenditure. There are no risks associated with this procedure.

D. Leeds Food Preference Questionnaire (LFPQ) (Approximately 15 minutes)-This task provides measures of the wanting and liking for an array of food images presented to participants on a computer screen. During the test, each food image is presented with every other food image in turn. Participants will be instructed to select the food you "most want to eat now" during each trial. Participants will also need to rate each of the visual food cues in turn on a 100-millimeter visual analogue scale (anchored by Not at all-Extremely), based on the following questions: "how much do you want some of this food now?" and "How pleasant would it be to experience a mouthful of this food now", respectively. This task will be completed at 60 minutes and 180 minutes post-breakfast consumption, immediately following lunch consumption.

E. Behavioral Choice Task - For this task, participants will sit in front of a laptop which will present to them 2 slot machine games: one is to earn points towards your preferred snack food and the other is to earn points towards your favorite fruit/vegetable. They will then have the opportunity to earn points towards your favorite snack and/or favorite fruit/vegetable by playing these different slot machines. To earn points, they must press a button on the mouse when the cursor is placed over the slot machine of choice, which then starts that slot machine. Points are then earned when all three objects on the screen match. This task will be completed immediately following the Leeds Food Preference Questionnaire administered at 180 minutes post-breakfast consumption and the amount of snack/ fruit earned during the game will be served with their lunch.

F. Olfactory (smell) capacity measurement -Participants will be required to complete 3 different odor tests. First, a set of 3 capsules will be subsequently presented to them and they must identify which of the 3 capsules presents an odor (the other 2 capsules are odorless). Second, a set of 3 capsules will be subsequently presented to them and them must identify which of the 3 capsules presents a different odor (the other 2 capsules will have the same odor). Finally, they will be required to identify the correct odor released by the capsule. Examples of some of the odors include rose, marker, banana, and grass.

G. Assessment of food intake at lunch (Approximately 30 minutes)-The energy intake of lunch will be measured with a test meal administered in the end of your experimental sessions (approximately 4 hours upon you arrive at the laboratory). This test meal will be selected from a food menu, which contains 57 different food and beverage items. Once the selected food items are prepared and served, participants will have 30 minutes to consume "as much or as little as they want" from the foods that you selected on the menu. The selected food items will then be prepared, measured and placed for you to eat at the lab.

Four follow-up sessions (approximately 90 minutes each) During the intervention, participants will be asked to visit the laboratory for a bi-weekly or a monthly evaluation (depending on the group to which you will be randomized). During these follow-up sessions we will evaluate participant's weight, resting metabolic rate and fasting appetite. As soon as they arrive at the laboratory (12 hours fasted), we will measure their current weight, appetite and resting metabolic rate. We will offer breakfast before participants leave. In total, participants will complete 3 follow-up visits.

FINAL EXPERIMENTAL SESSION (Approx. 6 hours) The same protocol applied at the baseline experimental session will be repeated after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Present a 30≥BMI≥40 kg/m2,
* Present a waist circumference >88 cm
* Must be weight-stable (±2 kg last 6 months)
* Must be sedentary (less than 150 minutes per week)
* Must be able to read in English
* Must to present no history of alcohol or drugs abuse
* Must be pre-menopausal with a regular menstrual cycle

Exclusion Criteria:

* present scores >12 in the 16-item Binge Score Symptoms and/or score >19 in the Depression Beck Inventory
* present any history or evidence of cardiovascular disease, peripheral vascular disease, or stroke;
* be insulin dependent (75g oral glucose tolerance test)
* present a known renal and/or liver disease
* present asthma requiring therapy
* present plasma cholesterol > 8 mmol/L
* present systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg
* present previous history of inflammation disease, or cancer,
* present untreated thyroid or pituitary disease
* consume regularly medications that could affect cardiovascular function and/or metabolism
* present food allergies
* be pregnant
* be smoker

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-01-02 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Resting energy expenditure after weight loss | 10 weeks
  Resting energy expenditure will be measured at baseline and in the end the intervention
Change in Resting energy expenditure after weight loss | 20 weeks
  Resting energy expenditure will be measured at baseline and in the end of the intervention

SECONDARY OUTCOMES:
Change in fasting Appetite sensations using a Visual Analogue scale after weight loss | 10 weeks
  appetite sensations using visual analogue scales will be measured in fasting state (12h) at baseline and in the end of the weight loss intervention
Change in fasting Appetite sensations using a Visual Analogue scale after weight loss | 10 weeks
  appetite sensations using visual analogue scales will be measured at 30,60,90,120,150,180min after breakfast at baseline and in the end of the weight loss intervention
Change in post-prandial Appetite sensations using a visual Analogue scale after weight loss | 20 weeks
  appetite sensations using visual analogue scales will be measured in fasting state (12h) at baseline and in the end of each intervention
Change in post-prandial Appetite sensations using a visual Analogue scale after weight loss | 20 weeks
  appetite sensations using visual analogue scales will be measured at 30,60,90,120,150,180min after breakfast at baseline and in the end of the weight loss intervention
changes in Food reward using the LFPQ after weight loss | 10 weeks
  explicit liking, explicit and implicit wanting will be measured using a tool called Leeds Preference Food Questionnaire. Measures will be taken at baseline and at the end of the intervention
changes in Food reward using the LFPQ after weight loss | 20 weeks
  explicit liking, explicit and implicit wanting will be measured using a tool called Leeds Preference Food Questionnaire. Measures will be taken at baseline and at the end of the intervention
changes in impulsivity using the Barrat Impulsiveness scale after weight loss | 10 weeks
  measures will be taken using a Barrat Impulsiveness scale at baseline and at the end of the intervention
changes in impulsivity using the Barrat Impulsiveness scale after weight loss | 20 weeks
  measures will be taken using a Barrat Impulsiveness scale at baseline and at the end of the intervention
changes in food reinforcement for favourite snack using a Behavioural choice task | 10 weeks
  food reinforcement will be measured using a Behavioural choice task, at 180 min after breakfast. Measures will be taken at baseline and at the end of the intervention.
changes in food reinforcement for favourite snack using a Behavioural choice computer task | 20 weeks
  food reinforcement will be measured using a Behavioural choice computer task at 180min after breakfast. Measures will be taken at baseline and at the end of the intervention.
changes in food reinforcement for favourite fruit using a Behavioural choice computer task | 10 weeks
  food reinforcement will be measured using a Behavioural choice computer task at 180min after breakfast. Measures will be taken at baseline and at the end of the intervention.
changes in food reinforcement for favourite fruit using a Behavioural computer choice task | 20 weeks
  food reinforcement will be measured using a Behavioural choice task at 180min after breakfast. Measures will be taken at baseline and at the end of the intervention.
changes in olfaction using the 'Sniffin Sticks' tests | 10 weeks
  Olfaction will be measured using the Sniffin' Sticks (Burghart Instruments, Wedel, Germany), a 3-test battery of odorized markers that measure odor detection threshold, odor discrimination, and odor identification at 90 min after breakfast at baseline and after intervention.
changes in olfaction using the 'Sniffin Sticks' tests | 20 weeks
  Olfaction will be measured using the Sniffin' Sticks (Burghart Instruments, Wedel, Germany), a 3-test battery of odorized markers that measure odor detection threshold, odor discrimination, and odor identification at 90 min after breakfast at baseline and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Doucet, PhD, Principal Investigator — Universiy of Ottawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hintze LJ, Doucet E, Goldfield GS. The relative reinforcing value of snack food is a significant predictor of fat loss in women with overweight or obesity. Appl Physiol Nutr Metab. 2022 Feb;47(2):134-140. doi: 10.1139/apnm-2021-0382. Epub 2021 Sep 27. PMID 34570984